CLINICAL TRIAL: NCT05594784
Title: Olverembatinib Combined With Reduced-Intensity Chemotherapy and Venetoclax for Newly Diagnosed Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia: A Prospective, Single-arm, Single-center Clinical Trial
Brief Title: Olverembatinib Combined With Reduced-Intensity Chemotherapy and Venetoclax for de Novo Ph+ ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022040
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-05

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
MeSH Terms: interventions — olverembatinib; venetoclax; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olverembatinib Combined With Reduced-Intensity Chemotherapy and Venetoclax (Experimental): For Induction cycle, olverembatinib will be given orally 40mg every other day. Patients with CMR, olverembatinib will be reduced to 30 mg every other day.
  Induction and consolidation cycles combined with a certain period of venetoclax.
  Reduced-intensity chemotherapy regimens consist mainly of vincristine and prednisone. Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT),or patients who keep BCR/ABL negative can receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation chemotherapy.
  Interventions: Drug: Olverembatinib; Drug: Venetoclax; Drug: prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: Olverembatinib — a third-generation TKI
Drug: Venetoclax — a selective inhibitor of B-cell lymphoma 2 (Bcl-2)
Drug: prednisone — Glucocorticoids
Drug: Vincristine — Anti-tumor alkaloids

SUMMARY:
The introduction of TKIs has greatly improved the prognosis of Ph+ ALL patients. The third-generation TKI ponatinib in combination with chemotherapy has demonstrated superior efficacy to first- and second-generation TKIs. However, unfortunately, ponatinib is not available in mainland China. Olverembatinib is the only third-generation TKI drug currently approved in mainland China. Venetoclax is an oral selective inhibitor of Bcl-2, and small exploratory clinical studies have demonstrated that venetoclax in combination with ponatinib showed high rates of CR as well as molecular response in relapsed/refractory Ph+ ALL. This study will explore the safety and efficacy of olverembatinib in combination with reduced-intensity chemotherapy and venetoclax in patients with newly diagnosed Ph+ ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 14 years or older
2. Newly diagnosed Philadelphia chromosome positive(either t(9;22) and/or BCR-ABL positive and/ or FISH positive) acute lymphoblastic leukemia; Patients will be diagnosed according to morphologic,immunologic, cytogenetic and molecular(MICM) criteria, including bone marrow morphology, immunophenotype, cytogenetic and molecular genetic (BCR/ABL gene, qualitative and quantitative analysis) examination
3. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
4. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤5 x ULN if leukemic involvement of the liver is present; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; normal electrolytes: Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN; Cardiac color Doppler ultrasound ejection fraction ≥ 45%;
5. Subject has provided written informed consent prior to any screening procedure

Exclusion Criteria:

1. Lymphoid blast crisis of chronic myelocytic leukemia (CML)
2. Previous or ongoing systemic anti-ALL therapy (including but not restricted to TKI and/or radiotherapy, except for appropriate pre-treatment)
3. Clinical manifestations of CNS or extramedullary involvement with ALL
4. Patients with a history of myocardial infarction within 12 months or clinically significant cardiac disorders disease (e.g., unstable angina, congestive heart failure, uncontrollable hypertension, uncontrollable arrhythmia, etc.)
5. Uncontrolled active serious infections that could, in the investigator's opinion, potentially interfere with the completion of treatment
6. Known HIV seropositivity
7. History of acute pancreatitis within 1 year of study screening or history of chronic pancreatitis
8. Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL)
9. Female patients who are pregnant or breast feeding
10. Poorly controlled diabetes, defined as glycosylated hemoglobin (HbA1c) values of >7.5%. Patients with preexisting, well-controlled diabetes are not excluded
11. Any serious psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
CMR rate | At 3 months of treatment (90 days)
  Complete molecular remission rate (CMR rate) at 3 months of treatment (90 days)

SECONDARY OUTCOMES:
Overall survival(OS) | up to 60 months
  From the date of registration to the date of death resulting from any cause
Relapse free survival | up to 60 months
  From the date of complete remission(CR) until the date of documented relapse or death due to any cause or the last follow-up day
The rate of adverse events | an expected average of 24 months
complete remission (CR) rate | an expected average of 3 months
The duration of CR | up to 60 months
The duration of molecular CR | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gong X, Liu W, Liu Y, Fang Q, Gu R, Liu K, Lin D, Zhou C, Zhang G, Gong B, Wei S, Li Y, Li S, Wang Y, Hu Y, Qiu S, Liu B, Wang Y, Mi Y, Wei H, Wang J. Olverembatinib combined with venetoclax and reduced-intensity chemotherapy for adult newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia: a single-center, single-arm, phase 2 trial. Leukemia. 2025 Aug;39(8):1838-1847. doi: 10.1038/s41375-025-02674-8. Epub 2025 Jun 30. PMID 40588568